CLINICAL TRIAL: NCT02303626
Title: OPuS-2: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Two Dose Levels of BCX4161 for 12 Weeks as an Oral Prophylaxis Treatment for Attacks of Hereditary Angioedema
Brief Title: 12-Week Safety and Efficacy Study of BCX4161 as an Oral Prophylaxis Against HAE Attacks
Acronym: OPuS-2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BCX4161-301
Record Dates: First submitted 2014-11-24; First posted 2014-12-01 (Estimated); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Hereditary Angioedema; HAE
Keywords: BCX4161; Prophylaxis; Prevention; HAE; Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — avoralstat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BCX4161 300 mg three times daily (Experimental): Three BCX4161 capsules (100 mg) and two placebo capsules to be taken three times daily by mouth
  Interventions: Drug: BCX4161; Drug: Placebo
- BCX4161 500 mg three times daily (Experimental): Five BCX4161 capsules (100 mg) to be taken three times daily by mouth
  Interventions: Drug: BCX4161
- Placebo three times daily (Placebo Comparator): Five placebo capsules to be taken three times daily by mouth
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BCX4161
  Arms: BCX4161 300 mg three times daily; BCX4161 500 mg three times daily
Drug: Placebo
  Arms: BCX4161 300 mg three times daily; Placebo three times daily

SUMMARY:
This study will evaluate the safety and efficacy of an oral treatment, BCX4161, in preventing acute attacks in participants with hereditary angioedema (HAE). Eligible participants will be randomized to receive one of two doses of BCX4161 or placebo for 12 weeks. The study will compare the number of acute attacks in each treatment group, as well as a number of other clinical outcomes, and the safety and tolerability of each dose of BCX4161 compared to placebo.

ELIGIBILITY:
Key Inclusion Criteria:

1. A clinical diagnosis of HAE type I or II
2. Documented HAE attacks within a defined calendar period; in the absence of documented HAE attacks, participants will be required to enter a run-in period to document attacks
3. Access to acute attack medications
4. Sexually active women of child-bearing potential and sexually active men must utilize highly effective contraception

Key Exclusion Criteria:

1. Women who are pregnant or breast-feeding
2. Any clinical condition or medical history that would interfere with the subject's safety or ability to participate in the study
3. Use of C1INH or tranexamic acid for prophylaxis of HAE attacks
4. Current participation in any other investigational drug study or within the last 30 days
5. History of or current alcohol or drug abuse
6. Infection with hepatitis B, hepatitis C or HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Riedl, MD MS, Principal Investigator — UCSD
Locations (39):
- United States (24):
  - Birmingham, Alabama
  - Scottsdale, Arizona
  - Granada Hills, California
  - San Diego, California
  - Walnut Creek, California
  - Colorado Springs, Colorado
  - Shreveport, Louisiana
  - Chevy Chase, Maryland
  - Boston, Massachusetts
  - Plymouth, Minnesota
  - St Louis, Missouri
  - New York, New York
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Lake Oswego, Oregon
  - Hershey, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
  - Galveston, Texas
  - Fairfax, Virginia
  - Spokane, Washington
  - Tacoma, Washington
- Leuven, Belgium
- Ottawa, Canada
- France (3):
  - Grenoble
  - Lille
  - Paris
- Germany (3):
  - Berlin
  - Frankfurt
  - Mörfelden-Walldorf
- Budapest, Hungary
- Milan, Italy
- United Kingdom (5):
  - Birmingham
  - Bristol
  - Cardiff
  - London
  - Manchester

REFERENCES:
- [Derived] Beard N, Frese M, Smertina E, Mere P, Katelaris C, Mills K. Interventions for the long-term prevention of hereditary angioedema attacks. Cochrane Database Syst Rev. 2022 Nov 3;11(11):CD013403. doi: 10.1002/14651858.CD013403.pub2. PMID 36326435

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from study sites in Belgium, Canada, France, Germany, Hungary, Italy, the United Kingdom and the United States, between December 2014 and October 2015
Groups:
- BCX4161 300 mg three times daily: Three BCX4161 capsules (100 mg) and two placebo capsules to be taken three times daily by mouth
  BCX4161
  Placebo
- BCX4161 500 mg three times daily: Five BCX4161 capsules (100 mg) to be taken three times daily by mouth
  BCX4161
- Placebo three times daily: Five placebo capsules to be taken three times daily by mouth
  Placebo
Period: Overall Study
Arm/Group | BCX4161 300 mg three times daily | BCX4161 500 mg three times daily | Placebo three times daily
Started | 36 | 38 | 36
Completed | 35 | 35 | 33
Not Completed | 1 | 3 | 3
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Subject Non-Compliance | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BCX4161 300 mg Three Times Daily | BCX4161 500 mg Three Times Daily | Placebo Three Times Daily | Total
Number analyzed (Participants) | 36 | 38 | 36 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (12.4) | 41.1 (15.1) | 42.1 (12.5) | 41.2 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 26 | 85
  Male | 7 | 8 | 10 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 0 | 0 | 0 | 0
  White | 32 | 36 | 34 | 102
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3 | 1 | 1 | 5
  Hungary | 1 | 1 | 4 | 6
  Belgium | 0 | 1 | 1 | 2
  United States | 19 | 19 | 17 | 55
  Italy | 1 | 4 | 0 | 5
  United Kingdom | 6 | 5 | 3 | 14
  France | 3 | 1 | 2 | 6
  Germany | 3 | 6 | 8 | 17
Qualifying attack rate [Mean (Standard Deviation); unit: Attacks/ week] — The study qualifying attack rate is based on run-in period attack rate or historical attack rate where historical attack data was not available. Run-in Attack Rate = Total Number of attacks reported during run - in period ∗ 7/ Duration of run-in period in days. Duration of run-in period is the date of the last qualifying attack - date of screening+1 and is reported in days. Historical Attack Rate =Total Number of Historical attacks reported ∗ 7/ Duration of historical reporting period in days. An HAE attack defined by pink rings on the skin/erythema marginatum.
  Attacks/ week | 0.93 (0.39) | 0.95 (0.39) | 0.92 (0.34) | 0.93 (0.37)

OUTCOME MEASURES:

1. Primary Outcome: The Mean Acute Angioedema Attack Rate
Description: An angioedema attack was defined as swelling at any location reported by participant, which had no swelling earlier. Total number of confirmed attacks during the treatment period standardized to a weekly attack-rate to adjust for the total duration of treatment. The attack rate was derived for each participant by treatment period. The weekly attack rate was equal to the total number of confirmed attacks during a treatment period divided by the duration of the treatment (in days) times 7 days.
Time Frame: 12 weeks
Population: The intent-to-treat (ITT) population included all participants who were randomized and received at least 1 dose of study intervention.
Measure: Least Squares Mean (Standard Error); unit: Confirmed attacks per week
Arm/Group | BCX4161 300 mg three times daily | BCX4161 500 mg three times daily | Placebo three times daily
Number analyzed (Participants) | 36 | 38 | 36
Confirmed attacks per week | 0.675 (0.089) | 0.589 (0.086) | 0.593 (0.088)

2. Secondary Outcome: Number of Attack-free Days
Description: The number of attack free days was the sum of the days during the treatment period for which participants reported no attacks.
Time Frame: 12 weeks
Population: The ITT population included all participants who were randomized and received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: Number of attack-free days
Arm/Group | BCX4161 300 mg three times daily | BCX4161 500 mg three times daily | Placebo three times daily
Number analyzed (Participants) | 36 | 38 | 36
Number of attack-free days | 62.8 (18.2) | 66.0 (17.9) | 63.6 (14.9)

3. Secondary Outcome: Number of Participants Who Are Attack-free
Description: The number of participants who reported no attacks during the 12-week treatment period.
Time Frame: 12 weeks
Population: The ITT population included all participants who were randomized and received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | BCX4161 300 mg three times daily | BCX4161 500 mg three times daily | Placebo three times daily
Number analyzed (Participants) | 36 | 38 | 36
Participants | 1 | 1 | 0

4. Secondary Outcome: Disease Activity, as Measured by the 84-day Angioedema Activity Score
Description: Angioedema Activity Score (AAS) consists of 5 questions (period in which swelling occurred, physical discomfort, daily activity restriction, cosmetic disfigurement, and overall severity) to be answered for each day during which a subject experiences an HAE attack. A score between 0 (no symptoms) and 3 (Severe symptoms) was assigned to the responses for each question and the total daily score will be derived as the sum of the 5 question scores for each day during which the subject experiences a confirmed attack. Daily AAS ranged from 0 to 15 with higher scores indicating the greater disease severity. For participants who completed the study, the 84-day AAS was obtained by sum of AAS score during the treatment period and ranged from 0 (best) to 1,260 (worst).For participants who discontinued the study prematurely the 84-day AAS was obtained using the formula: Sum of AAS score of each day on treatment ∗ 84/Number of days on treatment.
Time Frame: 12 weeks
Population: The ITT population included all participants who were randomized and received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BCX4161 300 mg three times daily | BCX4161 500 mg three times daily | Placebo three times daily
Number analyzed (Participants) | 36 | 38 | 36
score on a scale | 113.9 (101.9) | 88.5 (85.1) | 97.2 (77.3)

5. Secondary Outcome: Change From Baseline at Week 12, in Quality of Life as Measured by the Angioedema Quality of Life Questionnaire
Description: Angioedema Quality of Life questionnaire (AE-QoL) consisted of 4 domains (i.e., functioning, fatigue/mood, fear/shame, and nutrition) and a total score based on a total of 17 possible responses. The results of all the responses are summed up and transformed to a scale ranging from 0 (best) to 100 (worst).
Time Frame: Baseline (Day 1) and Week 12
Population: The ITT population included all participants who were randomized and received at least 1 dose of study intervention. Here 'Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BCX4161 300 mg three times daily | BCX4161 500 mg three times daily | Placebo three times daily
Number analyzed (Participants) | 33 | 36 | 33
score on a scale | -9.89 (3.11) | -17.45 (2.66) | -12.14 (2.64)

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant. No causal relationship with study drug or with the clinical study itself is implied. An AE could be an unfavorable and unintended sign, symptom (including an abnormal laboratory finding), syndrome, or illness that developed or worsened during the clinical study. A serious adverse event (SAE) is any untoward medical occurrence resulting in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, or other medically important event. Any graded abnormality that occurred following the initiation of study drug and up to 30 days after the last dose of study drug, and represented at least a 1-grade increase from the baseline assessment, was defined as treatment emergent.
Time Frame: From first dose up to 14 weeks
Population: The safety population included all randomized participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | BCX4161 300 mg three times daily | BCX4161 500 mg three times daily | Placebo three times daily
Number analyzed (Participants) | 36 | 38 | 36
Participants | 31 | 35 | 32

7. Secondary Outcome: Change From Baseline at Week 12 in Quality of Life, as Measured by the EuroQoL Five-dimensional, 5-level Questionnaire
Description: The EuroQoL five-dimensional, 5-level (EQ-5D-5L) was used to assess overall wellbeing and comprised the following five domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each domain has 5 response levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. It included the EQ Visual Analogue scale (EQ VAS) to rate overall health on a scale of 0 (worst health) to 100 (best health).
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BCX4161 300 mg three times daily | BCX4161 500 mg three times daily | Placebo three times daily
Number analyzed (Participants) | 34 | 36 | 32
score on a scale | 3.26 (2.38) | 2.41 (3.13) | 9.92 (1.72)

ADVERSE EVENTS:
Time Frame: From first dose up to 14 weeks.
Description: The safety population included all randomized participants who received at least 1 dose of study intervention.
Arm/Group | BCX4161 300 mg three times daily | BCX4161 500 mg three times daily | Placebo three times daily
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/38 | 0/36
Serious Adverse Events (participants affected / at risk) | 2/36 | 3/38 | 3/36
Other Adverse Events (participants affected / at risk) | 31/36 | 35/38 | 32/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCX4161 300 mg three times daily (N=36) | BCX4161 500 mg three times daily (N=38) | Placebo three times daily (N=36)
Hereditary angioedema (Congenital, familial and genetic disorders) | 2 (2) | 1 (1) | 1 (1) — HAE attack requiring hospitalization
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BCX4161 300 mg three times daily (N=36) | BCX4161 500 mg three times daily (N=38) | Placebo three times daily (N=36)
Abdominal distension (Gastrointestinal disorders) | 3 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 8 | 16 | 12
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1
Faeces soft (Gastrointestinal disorders) | 1 | 1 | 3
Flatulence (Gastrointestinal disorders) | 5 | 10 | 9
Frequent bowel movements (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 3 | 3
Hereditary angioedema (Congenital, familial and genetic disorders) | 2 | 1 | 1
Cystitis (Infections and infestations) | 1 | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 2
Influenza (Infections and infestations) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 5 | 8 | 7
Oral herpes (Infections and infestations) | 1 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 1 | 3
Tonsilitis (Infections and infestations) | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 2 | 1
Viral infection (Infections and infestations) | 1 | 2 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 0
Blood urine present (Investigations) | 3 | 0 | 0
GGT increased (Investigations) | 3 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 4 | 7 | 6
Somnolence (Nervous system disorders) | 0 | 1 | 2
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No